CLINICAL TRIAL: NCT06094582
Title: Knowledges and Use of Cannabidiol in Older Adults Aged 65 Years and Over in France
Brief Title: Knowledges and Use of Cannabidiol in Older Adults
Acronym: CBD-65
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0494; 2023-A02080-45 (Other: ID-RCB)
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aging; Frailty
Keywords: older adults; cannabidiol use; frailty
MeSH Terms: conditions — Frailty | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Participants will have to fulfill a short questionnaire (10 minutes) concerning their use and knowledges about CBD.

SUMMARY:
The use of non-medical cannabidiol (CBD) has been growing recently in France and in the world, in young but also older adults. Few data are available on the use of cannabidiol in older adults. A better knowledge of the use of cannabidiol in older adults, and of their own knowledges of the molecule, is necessary to guide and follow the CBD uptake in this population and avoid potential adverse events.

DETAILED DESCRIPTION:
Cannabidiol may be used by patients because it may have beneficial pharmacological effects (including anxiolytic, analgesic, anti-inflammatories or antioxidant effects). Older adults aged 65 years and over, are more frequently at risk of multimorbidity and loss of autonomy, and may present with several symptoms like pain, anxiety, sleep disturbances, that may potentially respond to CBD. The molecule is often marketed as devoid of adverse effects. Nevertheless, with ageing, reduction in liver and kidney function, may have an impact on the metabolism and elimination of CBD and increase the risk of side-effect. As well, the risk of interaction with drugs frequently prescribed in older adults such as CYP3A4 inhibitors (verapamil, ketoconazole …), CYP3A4 inducers (phenytoin, carbamazepine, …) or CY92C19 inhibitors or inducers (fluoxetine …), may increase the risk of side effects. Our hypothesis is that the use of CBD has increased last years in older adults, but that they are insufficiently informed about this molecule. There is a need to assess the prevalence of CBD use in older adults in France, to assess the knowledges of CBD users about this substance, and to better characterize CBD users.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the frailty clinic, in Toulouse University Hospital during the recruitment period.

Exclusion Criteria:

* major cognitive disorder with Mini Mental State Examination <20
* being under legal supervision or guardianship.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: older adults
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of CBD use (having consumed CBD at least once) | 1 day
  The patient will complete a questionnaire about CBD use

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine SOURDET, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France